CLINICAL TRIAL: NCT07194551
Title: Lynch Syndrome Carriers' Uterine Cancer Health Assessment: Sampling and DNA-based Detection
Brief Title: Assessing Uterine Cancer Risk in Lynch Syndrome Carriers Using Vaginal Self-sampling and a Health Questionnaire
Acronym: Lynch-SCAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other)
Responsible Party: Principal Investigator, Aline Talhouk, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: H24-00911
Record Dates: First submitted 2025-09-02; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Endometrial Cancer; Lynch Syndrome
Keywords: Reproductive Health; Lynch Syndrome
MeSH Terms: conditions — Endometrial Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaginal self-collection (Experimental): Participants will receive up to three at-home collection kits with a vaginal swab for DNA collection, a vaginal swab for microbiome sampling, a vaginal pH testing kit, and instructions on how to perform the sample collection. Vaginal DNA will be collected using Zymo DNA/RNA Shield, vaginal microbiome DNA will be collected using Genotek OMNIgene, and vaginal pH will be collected using GYNEX pHem-Alert.
  Participants with abnormal findings will be referred to a gynecologist or gynecologic oncologist for appropriate clinical assessment. Those with negative pathology will remain in the study. The self-collection will be repeated up to two more times, at eight-to-nine-month intervals, up to three successful self-collections.
  Interventions: Combination Product: Vaginal DNA swab, microbiome swab and pH test

INTERVENTIONS:
Combination Product: Vaginal DNA swab, microbiome swab and pH test — Participants will receive up to three at-home collection kits with a vaginal swab for DNA collection, a vaginal swab for microbiome sampling, a vaginal pH testing kit, and instructions on how to perform the sample collection. Vaginal DNA will be collected using Zymo DNA/RNA Shield, vaginal microbiome DNA will be collected using Genotek OMNIgene, and vaginal pH will be collected using GYNEX pHem-Alert. Those with abnormal findings will be referred to a gynecologist or gynecologic oncologist for appropriate clinical assessment. Those with negative pathology will remain in the study. The self-collection will be repeated up to two more times, at eight-to-nine-month intervals, up to three successful self-collections.
  Other Names: Zymo DNA/RNA Shield Swab Kit; DNAGenotek Inc. OMNIgene (OMR-130) Vaginal Microbiome Swab Kit; Gynex pHem-Alert Vaginal pH test

SUMMARY:
The goal of this study is to find out if self-collected vaginal swabs can be used to detect early signs of uterine cancer or related conditions in people with Lynch syndrome (LS) who still have their uterus. The study also tests if people with LS are willing and able to collect these samples themselves and whether they find the process acceptable.

The main questions this study asks are:

* Will people with LS take part in self-collection of vaginal samples, and do they find it acceptable?
* Can vaginal DNA mutations predict cancer risk or match results from other genetic or biopsy testing?
* Can a cancer risk model used in the general population also help identify risk in people with LS?

Participants will:

* Answer a health questionnaire about lifestyle and symptoms
* Collect their own vaginal swabs and measure their vaginal pH at home using a self-collection kit
* Complete short surveys around the time of self-collection and at the end of the study

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Lynch syndrome (confirmed by genetic testing).
* Have an intact uterus.
* Age 30 years or older.

Exclusion Criteria:

* History of endometrial cancer or endometrial hyperplasia.
* History of pelvic radiation or endometrial ablation.
* Pregnant at the time of study enrolment or during the study.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Acceptability of Self-collected Vaginal DNA to Assess for the Presence of Mutations Related to EC or EC Precursors | Through study completion, anticipated 1-2 years
  Feasibility will be measured by enrollment and adherence rates. Enrollment is defined as interested individuals completing the first round of self-collection. Adherence is defined as compliance with returning vaginal DNA samples, completing the health questionnaire, and submitting the exit survey. Acceptability will be measured through responses to a questionnaire post-self-collection and an exit survey, evaluating ease and overall experience with the self-collection process.

CONTACTS AND LOCATIONS:
Locations (1):
- VGH Research Pavilion, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No